CLINICAL TRIAL: NCT04867876
Title: Quality of Life Following Conservative Management for Pediatric Daytime Urinary Incontinence
Brief Title: Qol Following Management for Pediatric UI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Dakota (Other)
Responsible Party: Principal Investigator, Patti Berg-Poppe, Associate Professor, University of South Dakota
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QOL after UI treatment
Record Dates: First submitted 2015-01-06; First posted 2021-04-30 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2021-04

CONDITIONS: Quality of Life; Incontinence
Keywords: Quality of Life; Pediatric; Incontinence
MeSH Terms: interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention Cohort (Experimental): Physical Therapy
  Interventions: Behavioral: Physical Therapy

INTERVENTIONS:
Behavioral: Physical Therapy — Management of urinary incontinence by a physical therapist will include but is not limited to biofeedback, dietary management, alleviation of constipation, and neuromuscular re-education.

SUMMARY:
A comparison of changes between symptoms of incontinence and pediatric quality of life will be used to draw conclusions about whether differences in quality of life are noted with changes in symptoms of incontinence.

DETAILED DESCRIPTION:
Although positive physiological results are associated with successful treatment for bowel and bladder dysfunction and daytime incontinence (BD-UI), there are few studies examining the effects of treatment on quality of life (QoL) for children. The purpose of our study is to determine whether successful physical therapy treatment improves QoL for children with BD-UI.

Consent will be obtained from parents and assent from children. Children will be asked to complete a global, age appropriate quality of life assessment and a quality of life instrument specific to incontinence. Information will be provided by the parent through completion of a parent report instrument matched to the child's global quality of life tool as well as completion of an instrument depicting child symptoms. Clinicians will report general information about related physiological changes and progress with established outcomes individualized to the child. A repeated measures MANOVA will be used to analyze the results.

ELIGIBILITY:
Inclusion Criteria:

* Children between ages 5-18 who were currently receiving conservative treatment for daytime UI with or without constipation or encopresis met inclusion criteria.

Exclusion Criteria:

* Exclusion criteria included children who only had nocturnal enuresis or children with neurogenic bladders.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Dysfunctional Voiding Symptom Scale | 3-6 months
  Voiding dysfunction evaluation; scale 0-3; score of 8.5 or more is symptomology threshold
Kid KINDL Questionnaire | 3-6 months
  Quality of Life

CONTACTS AND LOCATIONS:
Overall Officials: Patti J. Berg-Poppe, PhD, Principal Investigator — University of South Dakota
Locations (1):
- University of South Dakota, Vermillion, South Dakota, United States